CLINICAL TRIAL: NCT06351228
Title: Outcomes of Early-stage Cervcial Cancer Patients Sheduled to Have Fertility-sparing Approach: The ETERNITY Project
Brief Title: Fertility-sparing in Early-stage Cervcial Cancer: The ETERNITY Project
Acronym: Eternity
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 5720
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Conization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Conization plus nodal evaluation — Conization plus nodal evaluation

SUMMARY:
The ETERNITY project is a retrospective analysis of outcomes of patients undergoing fertility-sparing treatment for cervcial cancer.

The primary aim is to report outcomes of those patients.

Other aims included:

1. Evaluation about the effectiveness of different treatment modalities;
2. Evaluation of outcomes according to different stages of disease;
3. Evaluation of the impactof neoadjuvant chemotherapy in patients undergoing conservative surgery

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed cervical cancer
* FIGO Stage IA1-IB3
* Fertility-sparing (conization plus nodal dissection)

Exclusion Criteria:

* age less than 18 yrs
* age more than 50 yrs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with early stage cervical cancer undegoing uterine preserving surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
oncological outcomes | 3-yrs
  disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bogani G, Scambia G, Malzoni M, Casarin J, Vizzielli G, Amant F, Raspagliesi F; Investigators of the ETERNITY Project. Chemo-conization in Early-sTage cERvical caNcer >2 cm scheduled for fertilItY-sparing approach: an analysis of the ETERNITY project. Int J Gynecol Cancer. 2025 Apr;35(4):101643. doi: 10.1016/j.ijgc.2025.101643. Epub 2025 Jan 17. PMID 39955179